CLINICAL TRIAL: NCT04036773
Title: The Impact of a Fruit and Vegetable Provision Program on Cardiovascular Health
Brief Title: Food Pharmacy at Oregon Health & Science University (OHSU) Knight Cardiovascular Institute (KCVI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Tracy Severson, dietitian, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19413
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Hyperlipidemias
Keywords: diet; nutrition; hyperlipidemia; produce
MeSH Terms: conditions — Hyperlipidemias | interventions — Fruit

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Dietary Supplement: Fruit and vegetable deliveries
- Control Group (No Intervention)

INTERVENTIONS:
Dietary Supplement: Fruit and vegetable deliveries — Weekly home deliveries of approximately 15 pounds of fresh fruits & vegetables
  Arms: Intervention Group

SUMMARY:
Participants in the intervention group of this study will receive weekly home deliveries of fruit & vegetables for 3 months. The primary objective of this study is to determine if increased access to fruits and vegetables leads to sustained dietary changes, measured through changes in the Healthy Eating Index (HEI). Secondary objectives are to determine whether increased fruit and vegetable access (increased HEI) ultimately leads to improved cardiovascular (CV) health indicators (e.g., body mass index, waist circumference, blood pressure, and levels of blood lipids and hemoglobin A1c).

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years and older
* Established patient at OHSU Center for Preventive Cardiology
* Not requiring changes to medication regimen for the 6-month study duration
* Must be eligible to register with produce delivery company (reside in Portland-metro area; have access to a computer with internet service; able to read English)

Exclusion Criteria:

* Triglycerides > 500 mg/dL
* Heavy alcohol use (> 3 drinks/day)
* Uncontrolled hypertension (BP > 140/90)
* LDL-C > 160 mg/dL
* Uncontrolled diabetes mellitus (HbA1c > 8%)
* Failure to provide informed consent
* Current pregnancy
* Healthy Eating Index (HEI) score of ≥ 80

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Intake of fruits and vegetables measured by changes in Healthy Eating Index (HEI) | 6 months
  The HEI uses a scoring system to evaluate a set of foods. The scores range from 0 to 100. An ideal overall HEI score of 100 reflects that the set of foods aligns with key dietary recommendations from the Dietary Guidelines for Americans.

SECONDARY OUTCOMES:
Changes in weight measured by body mass index | 6 months
  weight and height will be combined to report BMI in kg/m^2
Changes in waist circumference | 6 months
  Waist circumference will be measured in inches using a tape measure; desirable: < 40 inches (men), < 35 inches (women)
Changes in total cholesterol | 6 months
  measured via blood draw, desirable < 200 mg/dL
Changes in HDL-cholesterol | 6 months
  measured via blood draw, desirable > 40 mg/dL
Changes in LDL-cholesterol | 6 months
  measured via blood draw, desirable < 100 mg/dL
Changes in triglycerides | 6 months
  measured via blood draw, desirable < 150 mg/dL
Changes in blood pressure | 6 months
  Measured by medical assistant in clinic, desirable < 120/80 mmHg
Changes in blood glucose | 6 months
  measured via blood draw, desirable range is 60-99 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Severson, RDN, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No